CLINICAL TRIAL: NCT02315755
Title: OBSERVATIONAL STUDY EVALUATING THE EFFICACY OF TARGETED TREATMENTS FOLLOWING TYROSINE KINASE INHIBITORS IN METASTATIC RENAL CELL CARCINOMA PATIENTS AND EFFECTS ON QUALITY OF LIFE: A NATIONAL, MULTICENTER STUDY
Brief Title: Observational Study Evaluating The Efficacy And Effects On Quality Of Life Of Targeted Treatments Following TKIs In mRCC
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061086
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic renal cell carcinoma, targeted molecular therapy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study cohort: Metastatic renal cell carcinoma patients under 3rd line targeted therapy following 1st line interferon alpha and 2nd line TKI. All patients will be ≥ 18 years old and have signed the informed consent document.

SUMMARY:
Metastatic renal cell carcinoma (mRCC) is the most common malignant tumour of the kidneys. Targeted therapies, which were recently introduced in the treatment of mRCC, have become the standard treatment in these patients. With improved survival rate and a tolerable side effect profile, Tyrosine Kinase Inhibitors (TKIs) have largely replaced conventional immunotherapies worldwide.

In Turkey, due to reimbursement conditions, cytokine (interferon alpha) treatment is the standard treatment as first-line therapy.

Therefore, the data on quality of life (QoL) from the pivotal studies with standard TKI treatment does not reflect the QoL status of patients treated with TKIs as second or third line treatment in Turkey. In this study, the clinical outcomes and the impact on quality of life of targeted treatments following TKIs will be explored. To our knowledge, since there is no similar reimbursement condition in the world placing IFN as the first line standard treatment, this will be the first study evaluating the QoL status with targeted therapies used as 3rd line treatment in mRCC patients.

DETAILED DESCRIPTION:
Background:

Metastatic renal cell carcinoma (mRCC) is the most common malignant tumour of the kidneys. Targeted therapies, which were recently introduced in the treatment of mRCC, have become the standard treatment in these patients [1]. With improved survival rate and a tolerable side effect profile, Tyrosine Kinase Inhibitors (TKIs) have largely replaced conventional immunotherapies worldwide. [2-3] In Turkey, due to reimbursement conditions defined by the authority, cytokine (interferon alpha) treatment is the standard treatment as first-line therapy [4].

Rationale:

TKI therapy is used after interferon alpha in Turkey due to current reimbursement status. Therefore, the data on quality of life (QoL) from the pivotal studies with standard TKI treatment does not reflect the QoL status of patients treated with TKIs as second or third line treatment in Turkey. In this study, the clinical outcomes and the impact on quality of life of targeted treatments following TKIs will be explored. To our knowledge, since there is no similar reimbursement condition in the world placing IFN as the first line standard treatment, this will be the first study evaluating the QoL status with targeted therapies used as 3rd line treatment in mRCC patients.

Research Question and Objectives

Research Question:

There is no data available in the literature explaining the effect of targeted therapies used as 3rd line treatment following IFN and TKIs in metastatic renal cell carcinoma patients. Therefore, it is essential to understand health-related quality of life and efficacy of targeted therapies used as 3rd line treatment due to current reimbursement conditions in Turkey.

Primary Objective:

* Measurement of health-related quality of life with targeted therapy used as 3rd line treatment
* Overall response rate at the end of follow up
* Median progression free survival according to RECIST version 1.1

Secondary Objectives:

* Overall survival rate
* Effect of quality of life on prognosis.
* Adverse events during 3rd line targeted treatment according to CTCAE.4.03
* Dose modifications due to adverse events
* Correlation between efficacy (overall response rate at month 12 and median PFS) and dose modifications due to adverse events
* Correlation between efficacy (overall response rate at month 12 and median PFS) and blood pressure Study Design: This is a multi-center, national, non-interventional/observational study. It has been defined according to the NUTS (Nomenclature of Territorial Units for Statistics: Nomenclature d'unites Territoriales Statistiques, French) criteria, which is a regional classification, created in order to reduce interregional disparities in socio-economic analysis of the regions, and to produce data comparable to that of the European Union (EU). Turkey has been divided into 12 NUTS regions depending on the economic, social, cultural, and geographical aspects, and the population size. In this study, patients with metastatic renal cell carcinoma from centers in 12 NUTS regions of Turkey will be included, who meet the inclusion criteria. In this study, approximately 152 patients planned to be recruited in 12 months and followed-up for 12 months. Additionally, every patient will be followed-up once for survival follow-up in order to assess the overall survival before the site close out visit. Survival follow-up will be performed via telephone visit or site visit if exist.

Study Population:

Metastatic renal cell carcinoma patients under 3rd line targeted therapy following 1st line interferon alpha and 2nd line TKI. All patients will be ≥ 18 years old and have signed the informed consent document.

Variables:

Age, gender, height, weight, and vital signs such as blood pressure Socio-demographic characteristics ECOG performance status Concomitant diseases and medication Medical history Histopathological findings Type of the surgical procedure Treatment history and current treatment information Metastatic features MSKCC risk factors Laboratory findings The quality of life questionnaire (FKSI-15, EQ5D-3L, FKSI-DRS) on each visit. Blood pressure diary Other treatment during follow-up, if any, the dose and the duration Side effects (treatment of the side effects, interruption of the treatment, dose reduction, dose-elevation) PFS, OS and ORR evaluation during 3rd, 6th, 9th and 12th months performed according to RECIST version 1.1, additionally, every patient will be followed-up once for survival follow-up in order to assess the overall survival before the site close out visit. Survival follow-up will be performed via telephone visit or site visit if exist.

ORR: The best overall response is the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation. The patient's best overall response assignment will depend on the findings of both target and non-target disease and will also take into consideration the appearance of new lesions. Furthermore, depending on the nature of the study and the protocol requirements, it may also require confirmatory measurement.

PFS: The length of time during and after the treatment of a disease, that a patient lives with the disease but it does not get worse. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works.

OS: 1 year Overall Survival (OS), defined as the time from the start of 3rd line treatment until death or 1 year due to any cause (measured at the end of follow-up).

Data Sources: The source of the data will be the electronic or the written patient records of the participating centers. The patient's data can be accessed through a patient file. In the centers, both systems can be used in conjunction. The data can be accessed using both systems.

Sample Size: This is a multi-center, national, non-interventional/observational study. In this study, patients with metastatic renal cell carcinoma who meet the inclusion criteria will be included from centers in 12 NUTS regions of Turkey. Since this is a non-interventional observational study, there is no specific follow-up protocol. In this study, approximately 152 patients will be evaluated.

According to Turkish Statistical Institute data at the end of 2013 population of Turkey is approximately 80 million [5]. In the project of Turkey Association of Cancer Research Control which was named Cancer Record and Incidence shows that cancer incidence is 100-150 in 100.000 [6] and 2% of all new cancers are renal cell carcinoma [7]. There would be 1800 new RCC patients in 1 year, and according to the OS of the disease, there would be 4000 RCC patients in Turkey. 15% of these are metastatic at the time of diagnosis and 30-40% of these are metastatic after a period of a time [8]. Presuming that there are 1800 patients with metastatic renal carcinoma in Turkey, the minimum sample size with 7,6 confidence interval, 95% confidence level and 80% power was calculated as 152.

Data Analysis:

Statistical analyses will be primarily of explorative and descriptive nature. Patients who received at least one dose of 3rd line therapy and have sufficient information whether they had an adverse event or not will be valid for safety analysis. Patients who received at least one dose of 3rd line therapy and have any information regarding efficacy of therapy will be valid for intent-to-treat efficacy analysis.

Demographic data, baseline characteristics, diagnosis and prior treatment of RCC, concomitant diseases, and concomitant medication will be described with summary statistics such as mean, SD, minimum, 1, 5, 25, 75, 95, 99 percent quartiles, median, maximum for continuous variables, and category counts and frequencies (percentages) for categorical variables. Concomitant diseases on the case report form correspond to MedDRA terms. Concomitant medication will be coded using WHO's drug dictionary.

Descriptive summaries of Kaplan-Meier (KM) estimates (including number of failed, number censored, 25th and 75th percentiles with respective 95% confidence level and median with 95%Confidence level) and KM curves will be presented for time-to-event efficacy variables (PFS, TTP, time to treatment failure). Mean, SD, minimum, 1, 5, 25, 75, 95, 99 percent quartiles, median, maximum will be produced for duration of treatment. Category counts and frequencies (percentages) will be calculated for tumor status at different visits and general subjective rating of efficacy of 3rd line therapy from the treating physician.

Adverse events will be summarized using the CTCAE.4.03 coding system. Event rates for single adverse events will be calculated based on the total number of patients valid for safety. Adverse events will be categorized according to relation, seriousness, CTCAE grade (version 4.03), and discontinuation of therapy, action taken and outcome. Special attention will be paid to serious adverse events and unexpected or unlisted ADRs.

Category counts and frequencies (percentages) will be calculated for overall tolerability.

Since the enrollment is after the initiation of the treatment, some information will be collected and analyzed retrospectively.

The best overall response is the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation.

ELIGIBILITY:
Inclusion criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

* Histologically confirmed metastatic renal cell cancer patients who have already been using targeted therapies for up to 3 months as 3rd line treatment
* Patients older than 18 years
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legal representative) has been informed of all pertinent aspects of the study.

Exclusion criteria:

Patients meeting any of the following criteria will not be included in the study:

* Patients with contraindications for the use of the study medications
* Patients with (suspected) pregnancy or in lactation period
* Patients who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or patients who are Pfizer employees directly involved in the conduct of the trial.
* Participation in other studies involving investigational drug(s) (Phases 1-4) within 4 weeks before included in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic renal cell carcinoma patients under 3rd line targeted therapy following 1st line interferon alpha and 2nd line TKI. All patients will be ≥ 18 years old and have signed the informed consent document.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Turkey (Türkiye) (19):
  - Gazi University, Ankara, Besevler
  - Abdurrahman Yurtaslan Onkoloji Hastanesi, Ankara, Demetevler
  - Marmara Üniversitesi Pendik Eğtim Araştırma Hastanesi, Pendik, İ̇stanbul
  - Hacettepe University School of Medicine, Department of Medical Oncology, Ankara
  - Ankara Numune Egitim Arastirma Hastanesi, Ankara
  - Ege Universitesi Tip Fakultesi, Bornova/Izmir
  - Ali Osman Sonmez Onkoloji Hastanesi, Bursa
  - Dicle Universitesi Tip Fakultesi, Diyarbakır
  - Trakya Universitesi Tip Fakultesi Ic Hastaliklari Anabilim Dali Tibbi Onkoloji Bilim Dal, Edirne
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi Onkoloji Enstitusu, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Izmir Katip Celebi Universitesi Ataturk Egitim Arastirma Hastanesi Medikal Onkoloji Departmani, Izmir
  - Dr Lufti Kirdar Kartal Egitim ve Arastirma Hastanesi, Kartal
  - Konya Necmettin Erbakan Universitesi Meram Tip Fakultesi Tibbi Onkoloji Anabilim Dali, Konya
  - Inonu Universitesi Tip Fakultesi Medikal Onkoloji Bilim Dali, Malatya
  - Gaziantep Universitesi Tip Fakultesi, Sehitkamil/Gaziantep
  - Erciyes Universitesi Tip Fakultesi, Talas / Kayseri
  - Karadeniz Teknik Universitesi Tip Fakultesi Tibbi Onkoloji Bilim Dali, Trabzon

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061086&StudyName=Observational%20Study%20Evaluating%20The%20Efficacy%20Of%20Targeted%20Treatments%20Following%20Tyrosine%20Kinase%20Inhibitors%20In%20Metastatic%20Renal%20Cell%20Carcinoma%20Patients%20And%20Effects%20On%20Quality%20Of%20Life%3A%20A%20National%2C%20Multicenter%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Participants who had metastatic renal cell carcinoma and registered in centers of 12 Nomenclature of Territorial Units for Statistics (NUTS) regions of Turkey and met the inclusion criteria were observed in this study for 12 months. After 12 months, participants were followed up only once for survival follow up within the maximum study duration of 33 months.
Period: Overall Study
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Started | 102
Completed | 102 (Participants who died, were considered as 'completed'.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time duration (in months) during and after the treatment of disease that a participant lived with the disease but it did not get worse or progressed. Progressive disease as per response evaluation criteria in solid tumors (RECIST) version 1.1 defined as at least a 20 percent (%) increase in the sum of longest dimensions of target lesions, reference to the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions or increase of at least 5 millimeter (mm) in addition to the relative increase of 20%.
Time Frame: From the start of disease treatment until disease progression or death due to any cause (up to a maximum of 33 months)
Population: Analysis was performed on all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
months | NA [NA to NA] — Data was not estimable due to less number of participants with events.

2. Primary Outcome: Percentage of Participants With Overall Objective Response
Description: Overall objective response was defined as the percentage of participants with best confirmed response (partial response [PR], stable disease [SD] or progressive disease [PD]) recorded from the start of the study treatment until the end of treatment as assessed by RECIST version 1.1. PR defined as a 30% or more decrease in the sum of longest dimensions of the target lesions, taking as reference the baseline sum of longest dimensions. PD defined as at least a 20% increase in the sum of longest dimensions of target lesions, reference to the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions or increase of at least 5 mm in addition to the relative increase of 20%. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference to the smallest sum diameters while on study.
Time Frame: Baseline until the maximum of 33 months
Population: Analysis was performed on all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
percentage of participants
  PR | 23.5
  SD | 38.2
  PD | 18.6

3. Primary Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index - 15 (FKSI-15) Score at Baseline
Description: FKSI was used to assess quality of life (QoL) of the participants and consisted of 15 items (lack of energy, side effects, pain, losing weight, bone pain, fatigue, enjoying life, short of breath, worsened condition, appetite, coughing, bothered by fevers, ability to work, hematuria and sleep). Each of the 15 items was answered on a 5-point Likert scale ranging from 0 to 4 (0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, 4= very much). Total FKSI score = sum of the 15 item scores; total range: 0 - 60; 0 (no symptoms) to 60 (very much); higher score indicated greater presence of symptoms/worse quality of life.
Time Frame: Baseline (Day 1 of Month 1)
Population: Analysis was performed on all enrolled participants. Here, "overall number of participants analysed", indicates participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 99
units on a scale | 26 (6)

4. Primary Outcome: Change From Baseline in FKSI-15 Score at Month 3
Description: FKSI was used to assess QoL of the participants and consisted of 15 items (lack of energy, side effects, pain, losing weight, bone pain, fatigue, enjoying life, short of breath, worsened condition, appetite, coughing, bothered by fevers, ability to work, hematuria and sleep). Each of the 15 items was answered on a 5-point Likert scale ranging from 0 to 4 (0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, 4= very much). Total FKSI score = sum of the 15 item scores; total range: 0 - 60; 0 (no symptoms) to 60 (very much); higher score indicated greater presence of symptoms/worse quality of life.
Time Frame: Baseline (Day 1 of Month 1), Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 82
units on a scale | 1.2 (4.47)

5. Primary Outcome: Change From Baseline in FKSI-15 Score at Month 6
Description: as for outcome 3
Time Frame: Baseline (Day 1 of Month 1), Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 57
units on a scale | 1.21 (4.22)

6. Primary Outcome: Change From Baseline in FKSI-15 Score at Month 9
Description: as for outcome 3
Time Frame: Baseline (Day 1 of Month 1), Month 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 37
units on a scale | 1.38 (4.56)

7. Primary Outcome: Change From Baseline in FKSI-15 Score at Last Follow-up
Description: as for outcome 3
Time Frame: Baseline (Day 1 of Month 1), last follow-up visit (up to 33 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 30
units on a scale | 0.67 (5.27)

8. Primary Outcome: EuroQol-5 Dimension-3 Level (EQ5D-3L) Scores at Baseline
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions. Participants rated 5 aspects of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The mean of the summed score ranged from 1 to 3 with "1" corresponding to no problems and "3" corresponding to severe problems in the 5 dimensions, where higher score indicates more severe problems. Total index EQ-5D-3L summary score is weighted with a range of -0.594 (worst) to 1.0 (best).
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 100
units on a scale | 0.522 (0.236)

9. Primary Outcome: Change From Baseline in EQ5D-3L Scores at Month 3
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions. Participants rated 5 aspects of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The summed score ranged from 1-15 with "1" corresponding to no problems and "15" corresponding to severe problems in the 5 dimensions, where higher score indicates more severe problems.
Time Frame: Baseline (Day 1 of Month 1), Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 82
units on a scale | -0.07 (0.17)

10. Primary Outcome: Change From Baseline in EQ5D-3L Score at Month 6
Description: as for outcome 9
Time Frame: Baseline (Day 1 of Month 1), Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 57
units on a scale | -0.11 (0.34)

11. Primary Outcome: Change From Baseline in EQ5D-3L Score at Month 9
Description: as for outcome 9
Time Frame: Baseline (Day 1 of Month 1), Month 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 37
units on a scale | -0.06 (0.2)

12. Primary Outcome: Change From Baseline in EQ5D-3L Score at Last Follow-up
Description: as for outcome 9
Time Frame: Baseline (Day 1 of Month 1), last follow up visit (up to 33 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 30
units on a scale | -0.05 (0.39)

13. Primary Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index-Disease-Related Symptoms (FKSI-DRS) Score at Baseline
Description: FKSI-DRS was used to assess quality of life in participants and consisted of 9 items (lack of energy, pain, losing weight, bone pain, fatigue, short of breath, coughing, bothered by fevers, and hematuria). Each of the 9 items was answered on a 5-point Likert scale ranging from 0 to 4 (0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, 4= very much). Total FKSI-DRS score = sum of the 9 item scores; total range: 0 - 36; 0 (no symptom) to 36 (very much); higher score indicated greater presence of symptom.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 100
units on a scale | 14.56 (5.73)

14. Primary Outcome: Change From Baseline in FKSI-DRS Score at Month 3
Description: as for outcome 13
Time Frame: Baseline (Day 1 of Month 1), Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 82
units on a scale | 1.13 (3.81)

15. Primary Outcome: Change From Baseline in FKSI-DRS Score at Month 6
Description: as for outcome 13
Time Frame: Baseline (Day 1 of Month 1), Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 57
units on a scale | 1.04 (4.98)

16. Primary Outcome: Change From Baseline in FKSI-DRS Score at Month 9
Description: as for outcome 13
Time Frame: Baseline (Day 1 of Month 1), Month 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 37
units on a scale | 0.68 (4.94)

17. Primary Outcome: Change From Baseline in FKSI-DRS Score at Last Follow-up
Description: as for outcome 13
Time Frame: Baseline (Day 1 of Month 1), last follow up visit (up to 33 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 30
units on a scale | 1.6 (6.66)

18. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the start of 3rd line treatment until date of death due to any cause.
Time Frame: From the start of 3rd line treatment until death due to any cause (up to a maximum of 33 months)
Population: Analysis was performed on all enrolled participants.
Measure: Median (Full Range); unit: months
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
months | NA [NA to NA] — Data was not estimable due to less number of participants with events.

19. Secondary Outcome: Overall Survival at Year 1: Percentage of Participants Who Survived at Year 1
Description: Overall survival at Year 1 (Month 12) was defined as the time from the start of 3rd line treatment until death or 1 year due to any cause (measured at the end of 12 month follow-up/observation period). Percentage of participants who survived at the completion of 1 year (12 months) period were reported in this outcome measure.
Time Frame: Baseline until death due to any cause (up to 1 year)
Population: Analysis was performed on all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
percentage of participants | 79.9

20. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from the start of treatment to the date of disease progression or date of permanent discontinuation. PD as per RECIST version 1.1 was defined as at least a 20% increase in the sum of longest dimensions of target lesions, reference to the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions or increase of at least 5 mm in addition to the relative increase of 20%.
Time Frame: Baseline until disease progression or discontinuation, due to any cause (up to 33 months)
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 83
months | 4 [1 to 16]

21. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received disease treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant and jeopardized the participants or required treatment to prevent other AE outcomes for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment emergent AEs were events which occurred between start of disease treatment and up to Month 12 follow-up visit, that were absent before treatment or that worsened relative to pre-treatment state. AEs included both non-SAE and SAEs.
Time Frame: Baseline up to 12 months
Population: Analysis was performed on all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
Participants
  AEs | 33
  SAEs | 5

22. Secondary Outcome: Number of Participants With Grade 3 or Higher Severe Adverse Events (AEs) Based on NCI CTCAE Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received disease treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant and jeopardized the participants or required treatment to prevent other AE outcomes for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs were graded according to the National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 and coded using the Medical Dictionary for Regulatory Activities (MedDRA) as Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life threatening, Grade 5: Death related to AE. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 12 months
Population: Analysis was performed on all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
Participants | 13

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) During Third Line Targeted Treatment
Description: An AE was any untoward medical occurrence in a participant who received disease treatment without regard to possibility of causal relationship. Treatment emergent AEs during third line targeted treatment were events which occurred between first dose of third line targeted treatment and up to Month 12 follow-up visit, that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 12 months
Population: Analysis was performed on all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
Participants | 6

24. Secondary Outcome: Number of Participants With Dose Modifications of Third-Line Treatment Due to Adverse Events
Description: Number of participants that required dose modifications of third line treatment due to AEs were reported in this outcome measure. Dose modification was categorized as escalation (increase in dose), delay or interruptions (change in dose time or skipping any dose), reduction (decrease in dose).
Time Frame: Baseline up to Month 3, 6, 9 and 12
Population: Analysis was performed on all enrolled participants. Here, "Number analyzed, indicates participants evaluable for specified category".
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
Participants
  Escalation: Month 3: number analyzed (Participants) | 82
  Escalation: Month 3 | 7
  Interruption/delay: Month 3: number analyzed (Participants) | 82
  Interruption/delay: Month 3 | 13
  Reduction: Month 3: number analyzed (Participants) | 82
  Reduction: Month 3 | 4
  None: Month 3: number analyzed (Participants) | 82
  None: Month 3 | 58
  Escalation: Month 6: number analyzed (Participants) | 57
  Escalation: Month 6 | 5
  Interruption/delay: Month 6: number analyzed (Participants) | 57
  Interruption/delay: Month 6 | 7
  Reduction: Month 6: number analyzed (Participants) | 57
  Reduction: Month 6 | 2
  None: Month 6: number analyzed (Participants) | 57
  None: Month 6 | 43
  Escalation: Month 9: number analyzed (Participants) | 38
  Escalation: Month 9 | 0
  Interruption/delay: Month 9: number analyzed (Participants) | 38
  Interruption/delay: Month 9 | 5
  Reduction: Month 9: number analyzed (Participants) | 38
  Reduction: Month 9 | 0
  None: Month 9: number analyzed (Participants) | 38
  None: Month 9 | 33
  Escalation: Month 12: number analyzed (Participants) | 29
  Escalation: Month 12 | 0
  Interruption/delay: Month 12: number analyzed (Participants) | 29
  Interruption/delay: Month 12 | 4
  Reduction: Month 12: number analyzed (Participants) | 29
  Reduction: Month 12 | 0
  None: Month 12: number analyzed (Participants) | 29
  None: Month 12 | 25

25. Secondary Outcome: Correlation Coefficient Between Efficacy and Dose Modifications Due to AEs
Time Frame: Baseline up to Month 12 follow-up visit
Population: Analysis was performed on all enrolled participants.
Measure: Number; unit: Correlation coefficient
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
Correlation coefficient | NA — Data was not estimable due to less number of participants with dose modifications due to AEs.

26. Secondary Outcome: Correlation Coefficient Between Efficacy and High Blood Pressure (>150 / 90 Millimeter of Mercury )
Time Frame: Baseline up to Month 12 follow-up visit
Population: Analysis was performed on all enrolled participants.
Measure: Number; unit: Correlation coefficient
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 102
Correlation coefficient | NA — Data was not estimable due to less number of participants with High blood pressure.

ADVERSE EVENTS:
Time Frame: Baseline up to 12 months
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
All-Cause Mortality (participants affected / at risk) | 35/102
Serious Adverse Events (participants affected / at risk) | 5/102
Other Adverse Events (participants affected / at risk) | 33/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic Renal Cell Carcinoma (mRCC) Cohort (N=102)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mass in right on brochis (General disorders) | 1 — No vocabulary was used for this term and event.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic Renal Cell Carcinoma (mRCC) Cohort (N=102)
Diarrhoea (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 8
Hypertension (Vascular disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Angina pectoris (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Hypogonadism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pyrexia (General disorders) | 1
Swelling (General disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insomnia (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Cotton in mouth (General disorders) | 1 — No vocabulary was used for this term and event.
Inappetency (General disorders) | 2 — No vocabulary was used for this term and event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT02315755/Prot_SAP_000.pdf